CLINICAL TRIAL: NCT02054338
Title: Phase III Study of Vinflunine Plus Gemcitabine Versus Paclitaxel Plus Gemcitabine in Patients With Unresectable, Locally Recurrent or Metastatic Breast Cancer After Prior Anthracycline-based Adjuvant Chemotherapy
Brief Title: A Study of Vinflunine Plus Gemcitabine Versus Paclitaxel Plus Gemcitabine in Patients With Advanced Breast Cancer
Acronym: VICTORIA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was stopped before progressive disease or death of alive subjects.
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L00070 IN 303 B0; 2006-001139-23 (EudraCT Number)
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vinflunine plus gemcitabine (Experimental): vinflunine 320 mg/m² D1 plus gemcitabine 1000 mg/m2 D1 and D8 every 3 weeks
  Interventions: Drug: Vinflunine+Gemcitabine
- paclitaxel plus gemcitabine (Active Comparator): paclitaxel 175 mg/m² D1 followed by Gemcitabine 1250 mg/m² D1 and D8 every 3 weeks
  Interventions: Drug: Paclitaxel+Gemcitabine

INTERVENTIONS:
Drug: Vinflunine+Gemcitabine — Vinflunine 320 mg/m² IV on day 1 and.Gemcitabine 1000 mg/m² on days 1 and 8 of each cycle repeated every 3 weeks
  Other Names: L0070 IN
  Arms: vinflunine plus gemcitabine
Drug: Paclitaxel+Gemcitabine — paclitaxel 175 mg/m² on day 1 plus gemcitabine 1250 mg/m² on days 1
  Arms: paclitaxel plus gemcitabine

SUMMARY:
The combination of vinflunine and gemcitabine in advanced breast cancer in comparison to paclitaxel and gemcitabine is based on the following points: the significant antitumour activity of vinflunine in metastatic breast cancer (MBC) as single agent after anthracycline-taxane exposure and recent phase I study results of the vinflunine plus gemcitabine is at least additive and both drugs have a distinct mechanism of action; since taxanes have been approved in the adjuvant setting and are widely used in the treatment of early breast cancer it is worthwhile to assess new combination chemotherapy regimens as first line therapy for metastatic breast cancer.

DETAILED DESCRIPTION:
This is a randomised, multicentre, open-label phase III study comparing antitumour efficacy of vinflunine plus gemcitabine versus paclitaxel plus gemcitabine, as first line treatment for patients with unresectable, locally recurrent or metastatic breast cancer after prior anthracycline-based adjuvant chemotherapy.

Patients with metastatic breast cancer are incurable using conventional therapy with antitumoural hormonal drugs or cytostatic agents. The median survival from diagnosis of metastatic disease to death is reported to be approximately 3 years. While newer chemotherapeutic agents have been able to achieve tumour shrinkage, no significant increases in overall survival have been demonstrated so far. One reason for this result may be that breast cancer has a longer disease time span than NSCLC, allowing for administration of multiple therapies with different modalities. These therapies confound overall survival regardless of whether the treatment is a first-line or a subsequent treatment. The combination of gemcitabine plus paclitaxel has demonstrated improvement in overall survival over paclitaxel alone as first line therapy in patients with locally recurrent or metastatic breast cancer, however, this study compared single agent versus combination chemotherapy.

Using overall survival as a primary endpoint in a trial Using overall survival as a primary endpoint in a trial comparing 2 different cytostatic combinations in the treatment of metastatic breast cancer requires a large phase III study to detect a clinically significant difference. The advantages with such an endpoint are that it is technically easy to monitor and it is not dependent on monitoring tumour status. However, since patients with breast cancer typically receive 3 or more lines of chemotherapy, it becomes difficult to assess the impact of a first-line therapy on overall survival (as proposed herein) due to the potential for confounding effects from later treatments. A more specific instrument -if closely monitored- is progression-free survival. This endpoint reflects the impact of a specific treatment modality on the disease at a given time period and is probably confounded neither by prior treatments nor by subsequent therapies. Progression-free survival also represents an important clinical achievement for patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* 18 years or older but less than 75 years old
* histologically/cytologically confirmed breast cancer
* documented locally recurrent or metastatic breast cancer
* HER-2 negative or unknown
* prior neo- and/or adjuvant anthracycline-based chemotherapy
* measurable or non-measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.0
* adequate haematological, hepatic and renal functions
* ECG without any clinically relevant abnormality

Exclusion Criteria:

* known or clinical evidence of brain metastases or leptomeningeal involvement
* history of second primary malignancy
* patients having as sole tumour lesion: malignant effusion, lymphangitis, cystic lesion, bone lesion, and any other lesion not assessed by imaging techniques or colour photography
* pre-existing motor/sensory grade > 1 peripheral neuropathy
* prior therapy with vinca alkaloids and/or gemcitabine
* history of severe hypersensitivity to vinca alkaloids and/or gemcitabine or contraindication to any of these drugs
* pregnancy or breast feeding

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2006-06; Primary Completion 2011-06 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Keddad, MD, PhD, Study Director — Employed Pierre Fabre Medicament

RESULTS

PARTICIPANT FLOW:
Groups:
- Vinflunine Plus Gemcitabine: vinflunine 320 mg/m² D1 plus gemcitabine 1000 mg/m2 D1 and D8 every 3 weeks
  Vinflunine
  vinflunine plus gemcitabine: 320 mg/m² IV on day 1 plus gemcitabine 1000 mg/m² on days 1 and 8 of each cycle repeated every 3 weeks
- Paclitaxel Plus Gemcitabine: paclitaxel 175 mg/m² D1 followed by Gemcitabine 1250 mg/m² D1 and D8 every 3 weeks
  paclitaxel plus gemcitabine: paclitaxel 175 mg/m² on day 1 plus gemcitabine 1250 mg/m² on days 1
Period: Overall Study
Arm/Group | Vinflunine Plus Gemcitabine | Paclitaxel Plus Gemcitabine
Started | 503 | 501
Completed | 0 | 0
Not Completed | 503 | 501

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vinflunine Plus Gemcitabine | Paclitaxel Plus Gemcitabine | Total
Number analyzed (Participants) | 503 | 501 | 1004
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 428 | 438 | 866
  >=65 years | 75 | 63 | 138
Age, Continuous [Median (Full Range); unit: years] — The upper limit of full rage reported is higher than the one in the Eligibility Section of the Protocol. A total of 11 subjects (4 in the Vinflunine Plus Gemcitabine arm and 7 in the Paclitaxel Plus Gemcitabine arm) presented minor deviation at study entry.
  years | 53.2 [24.1 to 77.7] | 54.4 [21.5 to 79.0] | 53.6 [21.5 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 503 | 501 | 1004
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The primary efficacy parameter was Progression-free survival (PFS) analysed in the Intent-to-treat (ITT) population. PFS was defined as the time elapsed from randomisation date until the date of progression or death due to any cause (whichever came first).Tumor response was evaluated using the RECIST version 1.0 every 6 weeks until progression was recorded.
Time Frame: PFS was calculated from the registration date until the date of progression or death due to any cause if no progression was recorded first (median duration of follow-up: 14.1 months)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine Plus Gemcitabine | Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 503 | 501
Months | 8.0 [7.2 to 8.9] | 8.4 [7.6 to 8.9]
Statistical Analysis 1: Comparison: Vinflunine Plus Gemcitabine vs Paclitaxel Plus Gemcitabine; Kaplan-Meier curves and life tables by treatment arm to describe time-dependent parameters. Stratified Cox proportional model was used to compare the 2 treatment arms. A stratified Cox proportional hazards model and logistic regression were applied to the progression-free survival and to the tumour response, respectively; Test type: Superiority; p = 0.54, Log Rank; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.91 to 1.20]

2. Secondary Outcome: Overall Survival
Description: The secondary efficacy parameter was Overall Survival (OS) analysed in the Intent-to-treat (ITT) population. OS was defined as the time elapsed from the date of randomisation up to death or last follow-up.
Time Frame: OS was evaluated from the date of registration to the date of death due to any cause (median duration of follow-up: 14.1 months)
Population: ITT population - Cut-off date: 30 June 2011
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine Plus Gemcitabine | Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 503 | 501
Months | 18.9 [16.9 to 22.6] | 19.1 [17.8 to 21.4]
Statistical Analysis 1: Comparison: Vinflunine Plus Gemcitabine vs Paclitaxel Plus Gemcitabine; Test type: Superiority; p = 0.86, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.87 to 1.19]

3. Secondary Outcome: Overall Response Rate & Disease Control Rate
Description: Disease control rate (DCR) is defined as the sum of Complete Response (CR) and Partial Response (PR) and Stable Disease (SD) ≥ 6 months rate. Objective response rate (ORR) is defined as the sum of Complete Response (CR) and Partial Response (PR) rate (using the best confirmed response recorded from the date of randomisation to the end of treatment). DCR and ORR, assessed by Independent Review Committee using RECIST 1.0, were calculated in the ITT population.
Time Frame: ORR and DCR were calculated from the date of randomisation of first patient until the database cut-off (30 June 2011), assessed up to 5 years
Population: ITT
Measure: Median (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vinflunine Plus Gemcitabine | Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 503 | 501
percentage of patients
  Overall Response Rate | 11.3 [8.7 to 14.4] | 14.6 [11.6 to 18.0]
  Disease Control Rate | 39.8 [35.5 to 44.2] | 44.9 [40.5 to 49.4]
Statistical Analysis 1: Comparison: Vinflunine Plus Gemcitabine vs Paclitaxel Plus Gemcitabine; Test type: Superiority; p = 0.10, Log Rank; Hazard Ratio (HR) = 11.3, 95% CI 2-sided [8.7 to 14.4]

ADVERSE EVENTS:
Time Frame: Each subject was assessed for occurrence of Adverse Events throughout the study period (treatment period and follow-up period), up to 8 years.
Description: Safety data are presented for the global safety population which include the safety data of the 13 patients ongoing treatment (up to the premature termination date 18 February 2015). Safety population is defined as all treated patients analysed in the treatment arm they received (n=495 subjects in the Vinflunine Plus Gemcitabine arm and n=496 in the Paclitaxel Plus Gemcitabine arm)
Arm/Group | Vinflunine Plus Gemcitabine | Paclitaxel Plus Gemcitabine
All-Cause Mortality (participants affected / at risk) | 406/495 | 394/496
Serious Adverse Events (participants affected / at risk) | 215/495 | 128/496
Other Adverse Events (participants affected / at risk) | 494/495 | 494/496
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vinflunine Plus Gemcitabine (N=495) | Paclitaxel Plus Gemcitabine (N=496)
Anaemia (Blood and lymphatic system disorders) | 16 | 7 — Drug related
Febrile neutropenia (Blood and lymphatic system disorders) | 17 | 8 — Drug related
Leukopenia (Blood and lymphatic system disorders) | 7 | 3 — Drug related
Neutropenia (Blood and lymphatic system disorders) | 54 | 10 — Drug related
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 4 — Drug related
Atrial fibrillation (Cardiac disorders) | 3 | 2 — Drug related
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 — Drug related
Ventricular dysfunction (Cardiac disorders) | 1 | 0 — Drug related
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 — Drug related
Abdominal pain (Gastrointestinal disorders) | 19 | 1 — Drug related
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 — Drug related
Anal inflammation (Gastrointestinal disorders) | 1 | 0 — Drug related
Constipation (Gastrointestinal disorders) | 28 | 1 — Drug related
Diarrhoea (Gastrointestinal disorders) | 19 | 6 — Drug related
Dysphagia (Gastrointestinal disorders) | 2 | 0 — Drug related
Enterocolitis (Gastrointestinal disorders) | 2 | 0 — Drug related
Gastritis (Gastrointestinal disorders) | 0 | 1 — Drug related
Ileus (Gastrointestinal disorders) | 17 | 1 — Drug related
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 — Drug related
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1 — Drug related
Nausea (Gastrointestinal disorders) | 11 | 1 — Drug related
Odynophagia (Gastrointestinal disorders) | 1 | 0 — Drug related
Stomatitis (Gastrointestinal disorders) | 6 | 2 — Drug related
Vomiting (Gastrointestinal disorders) | 16 | 4 — Drug related
Asthenia (General disorders) | 2 | 3 — Drug related
Chest pain (General disorders) | 3 | 6 — Drug related
Condition aggravated (General disorders) | 5 | 3 — Drug related
Pyrexia (General disorders) | 11 | 13 — Drug related
Injection site reaction (General disorders) | 1 | 0 — Drug related
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 — Drug related
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 1 — Drug related
Anaphylactic reaction (Immune system disorders) | 0 | 1 — Drug related
Hypersensitivity (Immune system disorders) | 2 | 3 — Drug related
Bronchopneumonia (Infections and infestations) | 0 | 1 — Drug related
Catheter-related infection (Infections and infestations) | 5 | 2 — Drug related
Cellulitis (Infections and infestations) | 2 | 1 — Drug related
Erysipelas (Infections and infestations) | 2 | 1 — Drug related
Gastroenteritis (Infections and infestations) | 1 | 1 — Drug related
Infection NOS (Infections and infestations) | 0 | 2 — Drug related
Mastitis (Infections and infestations) | 0 | 1 — Drug related
Neutropenic infection (Infections and infestations) | 15 | 4 — Drug related
Neutropenic sepsis (Infections and infestations) | 1 | 0 — Drug related
Oral candidiasis (Infections and infestations) | 1 | 2 — Drug related
Orophrayngeal candidiasis (Infections and infestations) | 1 | 0 — Drug related
Pneumonia (Infections and infestations) | 10 | 13 — Drug related
Pyelonephritis (Infections and infestations) | 1 | 0 — Drug related
Sepsis (Infections and infestations) | 2 | 2 — Drug related
Septic shock (Infections and infestations) | 4 | 2 — Drug related
Soft tissue infection (Infections and infestations) | 1 | 0 — Drug related
Staphylococcal sepsis (Infections and infestations) | 0 | 1 — Drug related
Upper respiratory tract infection (Infections and infestations) | 0 | 1 — Drug related
Urinary tract infection (Infections and infestations) | 3 | 3 — Drug related
ALT increased (Investigations) | 1 | 1 — Drug related
AST increased (Investigations) | 1 | 1 — Drug related
Creatinine increased (Investigations) | 1 | 2 — Drug related
Transaminases increased (Investigations) | 2 | 1 — Drug related
Anorexia (Metabolism and nutrition disorders) | 5 | 5 — Drug related
Dehydration (Metabolism and nutrition disorders) | 11 | 2 — Drug related
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 — Drug related
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3 — Drug related
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 — Drug related
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 0 — Drug related
Hyponatraemia (Metabolism and nutrition disorders) | 13 | 0 — Drug related
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1 — Drug related
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 — Drug related
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 — Drug related
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — Drug related
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 — Drug related
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — Drug related
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 — Drug related
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 — Drug related
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Drug related
Encephalopathy (Nervous system disorders) | 1 | 0 — Drug related
Headache (Nervous system disorders) | 1 | 2 — Drug related
Paraesthesia (Nervous system disorders) | 2 | 0 — Drug related
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0 — Drug related
Syncope (Nervous system disorders) | 1 | 1 — Drug related
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Drug related
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 11 — Drug related
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Drug related
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 2 — Drug related
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Drug related
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 2 — Drug related
Pulmonary ooedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Drug related
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 2 — Drug related
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 — Drug related
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 — Drug related
Circulatory collapse (Vascular disorders) | 2 | 0 — Drug related
Embolism (Vascular disorders) | 0 | 1 — Drug related
Hypotension (Vascular disorders) | 4 | 3 — Drug related
Superior vena cava occlusion (Vascular disorders) | 0 | 2 — Drug related
Venous insufficiency (Vascular disorders) | 1 | 0 — Drug related
Fatigue (General disorders) | 17 | 5 — Drug related
Thrombocythamia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Generalized oedema (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 3 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Abscess soft tissue (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Genitourinary tract infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Nail bed infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 3
Tooth abscess (Infections and infestations) | 1 | 0
Viral pericarditis (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Bilirubin increased (Investigations) | 1 | 0
Hyperkaelemia (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 4 | 1
Depressed level of consciouness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic pulmonary obstructive disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Diabetes mellitus management (Surgical and medical procedures) | 0 | 1
Malignant tumour excision (Surgical and medical procedures) | 1 | 1
Deep venous thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypovolemic shock (Vascular disorders) | 0 | 1
Lymphooedema (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vinflunine Plus Gemcitabine (N=495) | Paclitaxel Plus Gemcitabine (N=496)
Anaemia (Blood and lymphatic system disorders) | 159 | 94 — Drug related
Leukopenia (Blood and lymphatic system disorders) | 34 | 27 — Drug related
Neutropenia (Blood and lymphatic system disorders) | 295 | 249 — Drug related
Thrombocytopenia (Blood and lymphatic system disorders) | 61 | 87 — Drug related
Abdominal pain (Gastrointestinal disorders) | 175 | 87 — Drug related
Abdominal pain upper (Gastrointestinal disorders) | 70 | 39 — Drug related
Constipation (Gastrointestinal disorders) | 239 | 126 — Drug related
Diarrhoea (Gastrointestinal disorders) | 111 | 137 — Drug related
Nausea (Gastrointestinal disorders) | 266 | 220 — Drug related
Stomatitis (Gastrointestinal disorders) | 169 | 85 — Drug related
Vomiting (Gastrointestinal disorders) | 216 | 134 — Drug related
Asthenia (General disorders) | 56 | 46 — Drug related
Fatigue (General disorders) | 314 | 286 — Drug related
Injection site reaction (General disorders) | 74 | 19 — Drug related
Oedema peripheral (General disorders) | 76 | 86 — Drug related
Pain (General disorders) | 49 | 40 — Drug related
Pyrexia (General disorders) | 124 | 133 — Drug related
Weight decreased (Investigations) | 166 | 126 — Drug related
Anorexia (Metabolism and nutrition disorders) | 164 | 119 — Drug related
Arthralgia (Musculoskeletal and connective tissue disorders) | 73 | 90 — Drug related
Bone pain (Musculoskeletal and connective tissue disorders) | 101 | 103 — Drug related
Myalgia (Musculoskeletal and connective tissue disorders) | 104 | 116 — Drug related
Pain in extremity (Musculoskeletal and connective tissue disorders) | 93 | 104 — Drug related
Dysgeusia (Nervous system disorders) | 19 | 34 — Drug related
Headache (Nervous system disorders) | 88 | 66 — Drug related
Paraesthesia (Nervous system disorders) | 22 | 75 — Drug related
Peripheral motor neuropathy (Nervous system disorders) | 11 | 34 — Drug related
Peripheral sensory neuropathy (Nervous system disorders) | 66 | 226 — Drug related
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 126 | 128 — Drug related
Alopecia (Skin and subcutaneous tissue disorders) | 202 | 317 — Drug related
Rash (Respiratory, thoracic and mediastinal disorders) | 39 | 65 — Drug related
Phlebitis (Vascular disorders) | 39 | 12 — Drug related
Febrile neutropenia (Blood and lymphatic system disorders) | 25 | 13
Dyspepsia (Gastrointestinal disorders) | 36 | 27
Chest pain (General disorders) | 57 | 49
Influenza like illness (General disorders) | 39 | 39
Upper respiratory tract infection (Infections and infestations) | 27 | 34
Urinary tract infection (Infections and infestations) | 37 | 37
Alanine aminotransferase increased (Investigations) | 25 | 27
Weight increased (Investigations) | 44 | 67
Dehydration (Metabolism and nutrition disorders) | 33 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 40 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 92 | 91
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 30 | 24
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 48 | 36
Dizziness (Nervous system disorders) | 25 | 27
Psychiatric disorders (Nervous system disorders) | 140 | 109
Anxiety (Nervous system disorders) | 51 | 46
Depression (Nervous system disorders) | 29 | 24
Insomnia (Nervous system disorders) | 81 | 57

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No